CLINICAL TRIAL: NCT01249144
Title: A Randomized Fellow-eye Controlled Clinical Trial to Compare the Visual and Refractive Outcomes Between Two Aspheric IOLs With Different Dioptric Increments and Manufacturing Tolerances in Patients Undergoing Bilateral Cataract Surgery
Brief Title: Visual and Refractive Outcomes After Implantation of Aspheric IOLs With Different Dioptric Increments and Manufacturing
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor stopped study to re-design trial
Sponsor: Lenstec Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTHD-10-05
Record Dates: First submitted 2010-11-24; First posted 2010-11-29 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2014-03

CONDITIONS: Cataract
Keywords: Intraocular Lens (IOL); Quarter Diopter; Biaspheric
MeSH Terms: conditions — Cataract | interventions — Lenses, Intraocular

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tecnis Z9002 Intraocular Lens (IOL) (Active Comparator)
  Interventions: Device: Intraocular Lens (IOL)
- Softec HD Intraocular Lens (IOL) (Active Comparator)
  Interventions: Device: Intraocular Lens (IOL)

INTERVENTIONS:
Device: Intraocular Lens (IOL) — Device for implantation in the capsular bag of the eye for visual correction of aphakia following cataract surgery.

SUMMARY:
This study compares two intraocular lenses, the Softec HD and the Tecnis Z9002, used to replace the natural crystalline lens after cataract extraction. The variables compared include 1) the accuracy of targeted versus achieved refractive outcomes and 2) visual acuity outcomes three months after implantation.

ELIGIBILITY:
Inclusion Criteria:

* operable cataracts in both eyes
* require intraocular lenses (IOLs) in dioptric range from 18.0 diopters to 25.0 diopters in both eyes
* </=1 diopter (D) of regular astigmatism in both eyes

Exclusion Criteria:

* Intraocular surgery or laser treatment prior to cataract surgery
* Severe dry eye
* Presence of ocular infection
* Uncontrolled intraocular pressure (IOP) or glaucoma preventing a postoperative best corrected visual acuity (BCVA) of 20/25 Snellen or better
* Retinal or macular pathology preventing a postoperative BCVA of 20/25 Snellen or better
* History of retinal detachment
* Corneal decompensation
* History of corneal disease (e.g., herpes simplex, herpes zoster keratitis, etc.)
* Clinically significant corneal endothelial dystrophy (e.g., Fuchs' dystrophy)
* Amblyopia preventing a postoperative BCVA of 20/25 Snellen or better

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Target versus Achieved Refraction | 3 Months Postoperative

SECONDARY OUTCOMES:
Uncorrected Visual Acuity | 3 Months Postoperative

CONTACTS AND LOCATIONS:
Overall Officials: J. Pitzer Gills, III, MD, Principal Investigator — St. Luke's Cataract and Laser Institute
Locations (1):
- St. Luke's Cataract & Laser Institute, Tarpon Springs, Florida, United States